CLINICAL TRIAL: NCT04520737
Title: Multimodal Prehabilitation During Neoadjuvant Chemotherapy in Patients With Colorectal Liver Metastases: a Randomized Controlled Trial
Brief Title: Multimodal Prehabilitation During Chemotherapy in Patients With Colorectal Liver Metastases
Acronym: PREHABMET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Responsible Party: Principal Investigator, Laia Estalella Mercade, Principal Investigator, Institut Investigacio Sanitaria Pere Virgili
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PREHABMET
Record Dates: First submitted 2020-08-11; First posted 2020-08-20 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Prehabilitation; Neoadjuvant Therapy; Liver Metastases
MeSH Terms: interventions — Psychosocial Intervention; Geriatric Assessment

STUDY DESIGN:
Intervention Model Description: The participant will be randomized (1:1) using seed, a Stata's random-number generated function. The subjects will be allocated into one of the two groups of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 16W group (Active Comparator): Multimodal prehabilitation program (MPP) will be implemented during 16 weeks, 12 weeks during chemotherapy (CT) and 4 weeks while waiting for surgery.
  Interventions: Behavioral: Physical Prehabilitation
- 4W group (Active Comparator): Multimodal prehabilitation program (MPP) will start at the end of preoperative chemotherapy (CT) until surgery (4 weeks in total).
  Interventions: Behavioral: Physical Prehabilitation

INTERVENTIONS:
Behavioral: Physical Prehabilitation — The prehabilitation program consists of the following interventions: in-hospital high-moderate intensive exercise training, nutritional assessment and high-protein supplementation, smoking cessation, psychological support and Comprehensive Geriatric Assessment.
  Other Names: Nutritional intervention; Psychological intervention; Smoking cessation; Comprehensive Geriatric Assessment (CGA) and co-morbidity assessment

SUMMARY:
Liver resection is the only curative treatment for patients with colorectal liver metastases (CRLM). Most patients undergo chemotherapy (CT) before liver surgery. CT objectively decreases patient functional capacity. It has already been demonstrated that a structured training program carried out during the 4 weeks following CT, while the patient is waiting for liver resection, is able to return the functional capacity to baseline levels. Despite this, multimodal prehabilitation programs (MPP) during preoperative CT have not been evaluated or implemented.

The aim of this study is to investigate whether a 16-week MPP applied during and following CT in CRLM patients will result in a significant increase in physical fitness when compared to those that undergo MPP only during the 4-weeks, between the end of CT and liver resection.

DETAILED DESCRIPTION:
The primary aim of the study is to evaluate the effectiveness of a multimodal prehabilitation program (MPP) in CRLM patients, which will be implemented right through the period of preoperative CT and during the 4-weeks of recovery before liver resection.

MPP will consist of in-hospital high-moderate intensive exercise training, nutritional assessment and high-protein supplementation, smoking cessation, psychological support and Comprehensive Geriatric Assessment.

Expected improvement in physical fitness will be measured by the difference in meters achieved in the six-minute walk test (6MWT) and will be compared with patients that will follow the MPP only during the 4-weeks before surgery, when preoperative CT has been finished.

Secondary aims include patient reported outcomes measures such as quality of life, postoperative complications, length of hospital stay, 30-day mortality and re-admissions. Protocol feasibility will be evaluated by monitoring all interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Written informed consent obtained from subject to participate in the study.

Exclusion Criteria:

* Age <18 years
* ASA health class status IV-V
* Mental conditions or disabling orthopedic and neuromuscular disease that prevent physical exercise or may compromise adherence to the program
* Medical contraindication to perform exercise
* Inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical Fitness- 6MWT | Baseline (before chemotherapy), week 12 (end of chemotherapy), week 16 (before surgery), 4 weeks postoperative, 8 weeks postoperative, 1 year postoperative
  Change in physical fitness will be measured by the six-minute walk test (6MWT). This test measures the distance an individual can walk, in metres, in a 6-minute period. Greater distance walked during the 6MWT indicates greater functional capacity.

SECONDARY OUTCOMES:
Postoperative complications- Clavien-Dindo classification | Through study completion, up to one year postoperative
  The Clavien-Dindo classification consists of 7 grades. Grade I: any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions; Grade II: Requiring pharmacological treatment with drugs other than such allowed for grade I complications; Grade III (IIIa, IIIb): Requiring surgical, endoscopic or radiological intervention; Grade IV (Iva, IVb): Life-threatening complication requiring IC/ICU management; Grade V: death of the patient.
Postoperative complications- CCI | Through study completion, up to one year postoperative
  The Comprehensive Complication Index (CCI) integrates in a single formula all complications by severity, ranging from 0 (uneventful course) to 100 (death).
Postoperative hospital length of stay | Postoperative period: assessed up to the first year postoperative
  The patient's postoperative length of stay will be recorded from the medical records. It will be calculated from the date of surgery until to the date of discharge from the hospital. It will be reported in days.
Readmissions rate | Postoperative period: Up to 30 postoperative days
  Rate of un-planned hospital readmissions within 30 days of discharge after hospitalization.
Functional capacity- 30CST | Baseline (before chemotherapy), week 12 (end of chemotherapy), week 16 (before surgery), 4 weeks postoperative, 8 weeks postoperative, 1 year postoperative
  The 30-second sit to stand test (30CST) measures lower body strength by recording the maximum number of times an individual can go from a seated position to a standing position, without using their arms, in a 30-second period.
Health-related quality of life- SF-36 | Baseline (before chemotherapy), week 16 (before surgery), 8 weeks postoperative, 1 year postoperative
  Quality of life will be evaluated by using the SF-36 mental health score. This survey measures eight scales of health: physical function, role physical, role emotional, social functioning, bodily pain, general health, vitality, and mental health. Each items are scored on a 0 to 100 range. A high score defines a more favorable health state.
Psychological health- HADS | Baseline (before chemotherapy), week 16 (before surgery), 8 weeks postoperative, 1 year postoperative
  Emotional health will be measured using the Hospital Anxiety and Depression Scale (HADS). The HADS contains seven items, each scored from 0 to 3 points for anxiety and depression. It provides summary measures on a scale of 0-21, with scores exceeding 8 suggesting the presence of a mood disorder
Functional capacity- Handgrip strength | Baseline (before chemotherapy), week 12 (end of chemotherapy), week 16 (before surgery), 4 weeks postoperative, 8 weeks postoperative, 1 year postoperative
  It will be measured using an hydraulic hand dynamometer. Three measures from each hand will be taken, with patient seated and arm bent at a 90-degree angle. The average of the three measures for each hand will be recorded.
Nutritional status- PG-SGA | Baseline (before chemotherapy), week 12 (end of chemotherapy), week 16 (before surgery), 4 weeks postoperative, 8 weeks postoperative, 1 year postoperative
  The Patient-Generated Subjective Global Assessment (PG-SGA) is a validated questionnaire used to assess the nutritional and functional status of cancer patients. The scoring system allows patients at risk for malnutrition to be identified and triaged for nutritional intervention. A score ≥9 indicates a critical need for nutritional intervention.
Nutritional status- BMI | Baseline (before chemotherapy), week 12 (end of chemotherapy), week 16 (before surgery), 4 weeks postoperative, 8 weeks postoperative, 1 year postoperative
  Body Mass Index (BMI) is weight in kilograms divided by height in meters squared.
Nutritional status- BIA | Baseline (before chemotherapy), week 12 (end of chemotherapy), week 16 (before surgery), 4 weeks postoperative, 8 weeks postoperative, 1 year postoperative
  The Bio-electrical Impedance Analysis (BIA) is a method to determine body composition. The measurement of body fat in relation to lean body mass.
Nutritional status- UMA | Baseline (before chemotherapy), week 12 (end of chemotherapy), week 16 (before surgery), 4 weeks postoperative, 8 weeks postoperative, 1 year postoperative
  Upper-arm muscle area (UMA) is the circumference of the left upper arm, measured at the mid-point between the tip of the shoulder and the tip of the elbow.

CONTACTS AND LOCATIONS:
Overall Officials: Laia Estalella, PhD, Principal Investigator — Hospital Universitari de Tarragona Joan XXIII
Locations (1):
- Hospital Universitari de Tarragona Joan XXIII, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No